CLINICAL TRIAL: NCT01486264
Title: An Open-Label, Non-Inferiority Study Evaluating the Efficacy and Safety of Two Injection Schedules of Xeomin® (incobotulinumtoxinA) [Short Flex Versus Long Flex] in Subjects With Cervical Dystonia With < 10 Weeks of Benefit From OnabotulinumtoxinA Treatment
Brief Title: Open-Label Non-Inferiority Study Evaluating the Efficacy and Safety of Xeomin® in Subjects With Cervical Dystonia Flex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Collaborators: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUS60201_4073_1
Record Dates: First submitted 2011-12-02; First posted 2011-12-06 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2017-04

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — incobotulinumtoxinA; Botulinum Toxins; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xeomin® Short Flex (Active Comparator): short flex dosing of Xeomin. It is a botulinum toxin type A produced from fermentation of Hall strain Clostridium botulinum serotype A.
  Interventions: Biological: Xeomin®
- Xeomin® Long Flex (Active Comparator): long flex dosing of Xeomin. It is a botulinum toxin type A produced from fermentation of Hall strain Clostridium botulinum serotype A.
  Interventions: Biological: Xeomin®

INTERVENTIONS:
Biological: Xeomin® — Xeomin is botulinum toxin type A produced from fermentation of Hall strain Clostridium botulinum serotype A
  Other Names: botulinum toxin; botulinum toxin type A

SUMMARY:
This study will compare Xeomin®, a botulinum toxin medication, in shorter treatment intervals (Short Flex dosing) to the standard interval dosing (Long Flex dosing) to determine if the response to treatment is comparable in both how it works and any side effects. Xeomin® is approved by the United States Food and Drug Administration (FDA) for the treatment of cervical dystonia (CD). The use of Xeomin® is investigational in regards to shorter treatment intervals. An investigational use is one that is not approved by the FDA.

DETAILED DESCRIPTION:
Dystonia is a movement disorder which is characterized by sustained, involuntary muscle contractions which frequently causes twisting and repetitive movements or abnormal postures of the trunk, neck, face, or arms and legs. In focal dystonia, the abnormal movements involve a single area of the body. A commonly described form of focal dystonia is cervical dystonia (CD). Botulinum toxin treatment can be offered as a treatment option for the treatment of CD.

The current practice for botulinum toxin injection treatment is to inject patients every 3 months. However, not all patients receive continuing benefit from botulinum toxin injections for an entire 3 months. In a recent survey, approximately 45% of patients report that they would prefer a treatment cycle of less than 10 weeks.This study will compare Xeomin®, a botulinum toxin treatment, in shorter treatment intervals (Short Flex dosing) to the standard interval dosing (Long Flex dosing) to determine if the response to treatment is comparable in both how it works and any side effects. Xeomin® is approved by the United States Food and Drug Administration (FDA) for the treatment of CD. The use of Xeomin® is investigational in regards to shorter treatment intervals. An investigational use is one that is not approved by the FDA.

The purpose of this research study is to evaluate the efficacy of the Short Flex dosing of Xeomin® compared to the Long Flex dosing regimen of Xeomin®, using a standard scale completed by the doctors and subjects as well as questionnaires that ask subjects to rate symptoms of CD.

ELIGIBILITY:
Inclusion Criteria:

* Documented clinical diagnosis of idiopathic or genetic Cervical Dystonia

Exclusion Criteria:

* Current treatment with botulinum toxin of any type for any other indication (including aesthetic indications) and for any body region during the study.

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2012-01-20 (Actual); Primary Completion 2016-03-29 (Actual); Study Completion 2016-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kulagowski, MD, Study Director — Merz North America, Inc.
Locations (43):
- United States (43):
  - Merz Investigative Site #001234, Birmingham, Alabama
  - Merz Investigative Site 001017, Fountain Valley, California
  - Merz Investigative Site #001225, Loma Linda, California
  - Merz Investigative Site #001219, Los Angeles, California
  - Merz Investigative Site # 001276, Manchester, Connecticut
  - Merz Investigative Site #001231, Washington D.C., District of Columbia
  - Merz Investigative Site #001076, Boca Raton, Florida
  - Merz Investigative Site #001019, Gainesville, Florida
  - Merz Investigative Site #001046, Jacksonville, Florida
  - Merz Investigative Site #001075, Melbourne, Florida
  - Merz Investigative Site #001217, Port Charlotte, Florida
  - Merz Investigative Site #1253, Tampa, Florida
  - Merz Investigative Site #001055, Atlanta, Georgia
  - Merz Investigative Site# 01255, Chicago, Illinois
  - Merz Investigative Site #001215, Chicago, Illinois
  - Merz Investigative Site # 01069, Des Moines, Iowa
  - Merz Investigative Site #001110, Overland Park, Kansas
  - Merz Investigative Site # 001071, Elkridge, Maryland
  - Merz Investigative Site # 001018, Detroit, Michigan
  - Merz Investigative Site #001030, Farmington Hills, Michigan
  - Merz Investigative Site # 0001275, Eagan, Minnesota
  - Merz Investigative Site #1250, St Louis, Missouri
  - Merz Investigative Site #001210, St Louis, Missouri
  - Merz Investigative Site #001221, Albany, New York
  - Merz Investigative Site #001233, New York, New York
  - Merz Investigative Site #1256, New York, New York
  - Merz Investigative Site# 01252, Charlotte, North Carolina
  - Merz Investigative Site #001005, Durham, North Carolina
  - Merz Investigative Site# 01260, Raleigh, North Carolina
  - Merz Investigative Site #001009, Winston-Salem, North Carolina
  - Merz Investigative Site #1265, Cincinnati, Ohio
  - Merz Investigative Site #001220, Tulsa, Oklahoma
  - Merz Investigative Site #1033, Portland, Oregon
  - Merz Investigative Site #1251, Portland, Oregon
  - Merz Investigative Site # 0001271, Hershey, Pennsylvania
  - Merz Investigative Site #1249, Philadelphia, Pennsylvania
  - Merz Investigative Site #001206, Nashville, Tennessee
  - Merz Investigative Site #1074, Dallas, Texas
  - Merz Investigative Site #001223, Dallas, Texas
  - Merz Investigative Site # 001216, Houston, Texas
  - Merz Investigative Site# 001266, Houston, Texas
  - Merz Investigative Site #001224, Kirkland, Washington
  - Merz Investigative Site #1270, Seattle, Washington

REFERENCES:
- [Result] Comella C, Hauser RA, Isaacson SH, Truong D, Oguh O, Hui J, Molho ES, Brodsky M, Furr-Stimming E, Comes G, Hast MA, Charles D. Efficacy and safety of two incobotulinumtoxinA injection intervals in cervical dystonia patients with inadequate benefit from standard injection intervals of botulinum toxin: Phase 4, open-label, randomized, noninferiority study. Clin Park Relat Disord. 2022 Mar 14;6:100142. doi: 10.1016/j.prdoa.2022.100142. eCollection 2022. PMID 35330880

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 43 sites in the United States.
Pre-assignment Details: A total of 283 participants were screened and randomized in the study. Of these, 282 participants were treated and 207 participants completed the study.
Groups:
- Xeomin Short Flex: Participants received Xeomin Short Flex, intramuscular injection, once on Day 1 (Visit 1) followed by 8 subsequent injection visits at 6 to 10 weeks interval for up to 762 days.
- Xeomin Long Flex: Participants received Xeomin Long Flex, intramuscular injection, once on Day 1 (Visit 1) followed by 8 subsequent injection visits at 90 days to 16 weeks interval for up to 875 days.
Period: Overall Study
Arm/Group | Xeomin Short Flex | Xeomin Long Flex
Started | 142 | 141
Treated | 142 | 140
Completed | 113 | 94
Not Completed | 29 | 47
Not completed — Death | 1 | 1
Not completed — Adverse Event | 3 | 3
Not completed — Lack of Efficacy | 6 | 10
Not completed — Withdrawal by Subject | 7 | 18
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 3 | 0
Not completed — Lost to Follow-up | 3 | 2
Not completed — Other | 5 | 11
Not completed — Not treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety evaluation set (SES) included all participants who were randomly assigned and received at least one study treatment, Xeomin Short-Flex or Long-Flex injection.
Groups:
- Total: Total of all reporting groups
Arm/Group | Xeomin Short Flex | Xeomin Long Flex | Total
Number analyzed (Participants) | 142 | 140 | 282
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (10.62) | 56.7 (11.30) | 57.1 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 98 | 204
  Male | 36 | 42 | 78
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 136 | 134 | 270
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 130 | 128 | 258
  Black or African American | 7 | 7 | 14
  Asian | 1 | 1 | 2
  American Indian or Alaska Native | 2 | 1 | 3
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  Other | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 142 | 140 | 282

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) Severity Subscale Score Based on Blinded Rater Assessment at Week 4 After the 8th Injection
Description: The validated assessment scale TWSTRS was used to measure the impact of cervical dystonia (CD) on participants. A blinded rater performed all TWSTRS-Severity subscale assessments for a given participant. TWSTRS-Severity subscale score ranges from 0 (=absence of severity) to 35 points (=maximum severity).
Time Frame: Baseline and Week 4 after the 8th injection (Week 44 to 68 for Short Flex and Week 84 to 104 for Long Flex)
Population: The per protocol set (PPS) included all participants in the full analysis set (FAS) who was responsive to unilateral brow injection (UBI) at the 4-week control visit after initial injection or had no major protocol deviations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Xeomin Short Flex | Xeomin Long Flex
Number analyzed (Participants) | 101 | 79
score on a scale | -4.1 (5.5) | -2.4 (5.4)
Statistical Analysis 1: Comparison: Xeomin Short Flex vs Xeomin Long Flex; Test type: Non-Inferiority — Analysis of covariance (ANCOVA) model adjusted for the baseline TWSTRS Severity subscale score, was used to test the non-inferiority of Short Flex versus Long Flex treatment. Non-inferiority margin delta equal to (=) 2 points; Least Square (LS) Mean difference = -1.4, 95% CI 2-sided [-2.9 to 0.1], Standard Error of Mean 0.75

2. Secondary Outcome: Change From Baseline in TWSTRS Total Score Based on Blinded Rater Assessment at Week 4 After the 8th Injection
Description: The validated assessment scale TWSTRS was used to measure the impact of CD on participants. The scale comprised of 3 subscales: Severity, Disability, and Pain, each of which was scored independently. A blinded rater performed all TWSTRS assessments for a given participant. TWSTRS-Severity subscale score ranges from 0 (=absence of severity) to 35 points (=maximum severity); TWSTRS-Disability subscale score ranges from 0 (no disability) to 30 (maximum disability); and TWSTRS-Pain subscale score ranges from 0 (no pain) to 20 (maximum pain). The total of these 3 comprises the TWSTRS total score which is scored from 0 (no symptoms) to 85 (worst symptoms). Higher scores indicate a greater impact of CD on participant.
Time Frame: Baseline and Week 4 after the 8th injection (Week 44 to 68 for Short Flex and Week 84 to 104 for Long Flex)
Population: FAS was subset of SES participants who were randomly assigned and received at least one injection and for whom TWSTR-Severity value by a blinded rater was available at baseline injection visit and control visit 4 weeks after the 8th injection. Participants who were evaluable for this measure at a given time point were included for this assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Xeomin Short Flex | Xeomin Long Flex
Number analyzed (Participants) | 101 | 79
score on a scale | -8.5 (10.3) | -7.6 (11.0)

3. Secondary Outcome: Change From Baseline in TWSTRS Total Score Based on Unblinded Rater Assessment at Week 4 After the 8th Injection
Description: The validated assessment scale TWSTRS was used to measure the impact of CD on participant. The scale comprised of 3 subscales: Severity, Disability, and Pain, each of which was scored independently. An unblinded rater performed all TWSTRS assessments for a given participant. TWSTRS-Severity subscale score ranges from 0 (=absence of severity) to 35 points (=maximum severity); TWSTRS-Disability subscale score ranges from 0 (no disability) to 30 (maximum disability); and TWSTRS-Pain subscale score ranges from 0 (no pain) to 20 (maximum pain). The total of these 3 comprises the TWSTRS total score which is scored from 0 (least symptoms) to 85 (worst symptoms). Higher scores indicate a greater impact of CD on participant.
Time Frame: Baseline and Week 4 after the 8th injection (Week 44 to 68 for Short Flex and Week 84 to 104 for Long Flex)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Xeomin Short Flex | Xeomin Long Flex
Number analyzed (Participants) | 101 | 79
score on a scale | -9.4 (11.1) | -10.3 (10.9)

4. Secondary Outcome: Change From Baseline in TWSTRS Severity Subscale Based on Unblinded Rater Assessment at Week 4 After the 8th Injection
Description: The validated assessment scale TWSTRS was used to measure the impact of cervical dystonia (CD) on participants. An unblinded rater performed all TWSTRS-Severity subscale assessments for a given participant. TWSTRS-Severity score ranges from 0 (absence of severity) to 35 (maximum severity).
Time Frame: Baseline and Week 4 after the 8th injection (Week 44 to 68 for Short Flex and Week 84 to 104 for Long Flex)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Xeomin Short Flex | Xeomin Long Flex
Number analyzed (Participants) | 101 | 79
score on a scale | -4.8 (6.2) | -5.1 (4.9)

5. Secondary Outcome: Change From Baseline in TWSTRS Disability Subscale Based on Unblinded Rater Assessment at Week 4 After the 8th Injection
Description: The validated assessment scale TWSTRS was used to measure the impact of CD on participant. An unblinded rater performed all TWSTRS-Disability subscale assessments for a given participant. TWSTRS-Disability score ranges from 0 (no disability) to 30 (maximum disability).
Time Frame: Baseline and Week 4 after the 8th injection (Week 44 to 68 for Short Flex and Week 84 to 104 for Long Flex)
Population: The FAS was the subset of the SES participants who were randomly assigned and received at least one injection and for whom a TWSTR-Severity value by a blinded rater (primary variable) was available at the baseline injection visit and the control visit 4 weeks after the 8th injection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Xeomin Short Flex | Xeomin Long Flex
Number analyzed (Participants) | 108 | 90
score on a scale | -1.9 (4.5) | -2.1 (5.8)

6. Secondary Outcome: Change From Baseline in TWSTRS Pain Subscale Based on Unblinded Rater Assessment at Week 4 After the 8th Injection
Description: The validated assessment scale TWSTRS was used to measure the impact of CD on participants. An unblinded rater performed all TWSTRS-Pain subscale assessments for a given participant. TWSTRS-Pain score ranges from 0 (no pain) to 20 (maximum pain).
Time Frame: Baseline and Week 4 after the 8th injection (Week 44 to 68 for Short Flex and Week 84 to 104 for Long Flex)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Xeomin Short Flex | Xeomin Long Flex
Number analyzed (Participants) | 108 | 90
score on a scale | -2.7 (4.2) | -3.1 (4.9)

7. Secondary Outcome: Change From Control Visit Week 4 After First Injection in Investigator-Rated Global Response at Week 4 After the 8th Injection
Description: The Investigator-Rated Global Response assessment for each Xeomin treatment was scored using a 9-point scale with a score ranging from -4 to +4 as follows: -4 (very marked worsening); -3 (marked worsening); -2 (moderately worsening); 1 (minimally worsening); 0 (no change); +1 (minimally improved); +2 (moderately improved); +3 (significantly improved); +4 (complete abolishment of signs and symptoms).
Time Frame: Week 4 and Week 4 after the 8th injection (Week 44 to 68 for Short Flex and Week 84 to 104 for Long Flex)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Xeomin Short Flex | Xeomin Long Flex
Number analyzed (Participants) | 104 | 90
score on a scale | -0.3 (1.47) | -0.1 (1.45)

8. Secondary Outcome: Change From Control Visit Week 4 After First Injection in Subject-Rated Global Response at Week 4 After the 8th Injection
Description: The Subject-Rated Global Response assessment for each Xeomin treatment was scored using a 9-point scale with a score ranging from -4 to +4 as follows: -4 (very marked worsening); -3 (marked worsening); -2 (moderately worsening); 1 (minimally worsening); 0 (no change); +1 (minimally improved); +2 (moderately improved); +3 (significantly improved); +4 (complete abolishment of signs and symptoms).
Time Frame: Week 4 and Week 4 after the 8th injection (Week 44 to 68 for Short Flex and Week 84 to 104 for Long Flex)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Xeomin Short Flex | Xeomin Long Flex
Number analyzed (Participants) | 103 | 90
score on a scale | 0.4 (1.61) | 0.5 (1.79)

9. Secondary Outcome: Change From Control Visit Week 4 After First Injection in Subject Satisfaction Score at Week 4 After the 8th Injection
Description: The Subject Satisfaction assessment for each Xeomin treatment was scored using a 10-point scale to answer the question, "How satisfied are you at the moment with your current therapy? Score ranges from: 1 (completely satisfied) to 10 (completely unsatisfied).
Time Frame: Week 4 and Week 4 after the 8th injection (Week 44 to 68 for Short Flex and Week 84 to 104 for Long Flex)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Xeomin Short Flex | Xeomin Long Flex
Number analyzed (Participants) | 94 | 89
score on a scale | -1.2 (3.42) | -0.6 (3.42)

10. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity
Description: Assessment of Clinical Global Impression Severity was scored using a 7-point scale for severity of illness, in response to the question, "Considering your total clinical experience with this particular population, how ill is the participant at this time?" With scores as: 0 (not assessed); 1 (normal, not ill at all); 2 (borderline ill); 3 (mildly ill); 4 (moderately ill); 5 (markedly ill); 6 (severely ill); and 7 (among the most extremely ill participants).
Time Frame: Baseline and 8th injection (Week 44 for Short Flex and Week 84 for Long Flex)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Xeomin Short Flex | Xeomin Long Flex
Number analyzed (Participants) | 107 | 90
score on a scale | -0.5 (0.89) | -0.1 (1.03)

11. Secondary Outcome: Change From Baseline in Cervical Dystonia Impact Profile-58 (CDIP-58) Total Score at Week 4 After the 8th Injection
Description: The CDIP-58 assesses the health impact of CD. The CDIP-58 is composed of eight domains: head and neck (6 items; 6 to 30 points), pain and discomfort (5 items; 5 to 25 points), upper limb activities (9 items; 9 to 45 points), walking (9 items; 9 to 45 points), sleep (4 items; 4 to 20 points), annoyance (8 items; 8 to 40 points), mood (7 items; 7 to 35 points), and psychosocial functioning (10 items; 10 to 50 points). Subscale scores were transformed to a common theoretical range of 0 (no impact) to 100 (most impact). Transformation to a 0 to 100 scale for the sum scores of the sub- and total scales were done using the following formula (all single items have scores from 1 to 5): S0 to 100 =25 * ([ SO / NI] - 1), S0 to 100 = transformed sum score. SO = sum score of the original sub- / total scale. NI = number of items in the sub- / total scale. Negative changes from the baseline total score indicate improvement in the impact of CD on health whereas positive changes indicate worsening.
Time Frame: Baseline and Week 4 after the 8th injection (Week 44 to 68 for Short Flex and Week 84 to 104 for Long Flex)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Xeomin Short Flex | Xeomin Long Flex
Number analyzed (Participants) | 108 | 90
score on a scale | -14.42 (20.377) | -12.45 (18.457)

12. Secondary Outcome: Change From Baseline in CDIP-58 Subscales' Scores at Week 4 After the 8th Injection
Description: The CDIP-58 assesses the health impact of CD. The CDIP-58 is composed of eight domains: head and neck (6 items; 6 to 30 points), pain and discomfort (5 items; 5 to 25 points), upper limb activities (9 items; 9 to 45 points), walking (9 items; 9 to 45 points), sleep (4 items; 4 to 20 points), annoyance (8 items; 8 to 40 points), mood (7 items; 7 to 35 points), and psychosocial functioning (10 items; 10 to 50 points). Subscale scores were transformed to a common theoretical range of 0 (no impact) to 100 (most impact). Negative changes from the baseline scores indicate improvement in the impact of CD on health whereas positive changes indicate worsening.
Time Frame: Baseline and Week 4 after the 8th injection (Week 44 to 68 for Short Flex and Week 84 to 104 for Long Flex)
Population: The FAS was the subset of the SES who were randomly assigned and received at least one injection and for whom a TWSTR-Severity value by a blinded rater (primary variable) was available at the baseline injection visit and the control visit 4 weeks after the 8th injection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Xeomin Short Flex | Xeomin Long Flex
Number analyzed (Participants) | 108 | 90
score on a scale
  Head and neck score | -22.49 (24.699) | -23.70 (27.152)
  Pain and discomfort score | -13.79 (27.912) | -7.92 (23.906)
  Sleep score | -12.79 (29.045) | -9.97 (26.158)
  Upper limb activities score | -8.98 (22.822) | -8.27 (20.982)
  Walking score | 8.41 (809) | -7.01 (20.884)
  Annoyance score | 15.83 (25.735) | -9.69 (24.771)
  Mood score | -14.52 (24.307) | -10.20 (23.137)
  Psychosocial functioning score | -15.90 (24.764) | -15.81 (23.428)

13. Secondary Outcome: Time to Offset of Xeomin Effects by Injection Cycle
Description: The Offset Questionnaire was a single question: "On most days last week, have you noticed that your CD symptoms are better, worse or the same as the week prior? Time to offset of effect was calculated from date of first onset of effect to date of offset of effects.
Time Frame: Week 4 up to Week 112
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Xeomin Short Flex | Xeomin Long Flex
Number analyzed (Participants) | 108 | 90
weeks
  Injection 1: number analyzed (Participants) | 69 | 49
  Injection 1 | 4.8 (2.85) | 5.8 (3.89)
  Injection 2: number analyzed (Participants) | 66 | 47
  Injection 2 | 4.8 (2.60) | 6.8 (3.83)
  Injection 3: number analyzed (Participants) | 58 | 50
  Injection 3 | 5.0 (2.31) | 7.8 (3.52)
  Injection 4: number analyzed (Participants) | 54 | 45
  Injection 4 | 5.1 (2.60) | 8.6 (3.70)
  Injection 5: number analyzed (Participants) | 47 | 43
  Injection 5 | 5.4 (3.00) | 9.2 (3.05)
  Injection 6: number analyzed (Participants) | 45 | 33
  Injection 6 | 6.4 (2.36) | 9.5 (2.50)
  Injection 7: number analyzed (Participants) | 35 | 32
  Injection 7 | 5.4 (2.63) | 9.1 (2.80)
  Injection 8: number analyzed (Participants) | 12 | 0
  Injection 8 | 4.2 (1.94) |

ADVERSE EVENTS:
Time Frame: Baseline up to Day 875
Description: The investigator asked the participant for adverse events (AEs) systematically at each visit.
Arm/Group | Xeomin Short Flex | Xeomin Long Flex
All-Cause Mortality (participants affected / at risk) | 1/142 | 1/140
Serious Adverse Events (participants affected / at risk) | 15/142 | 11/140
Other Adverse Events (participants affected / at risk) | 77/142 | 77/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Xeomin Short Flex (N=142) | Xeomin Long Flex (N=140)
Pneumonia (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Syncope (Nervous system disorders) | 2 | 0
Burning sensation (Nervous system disorders) | 0 | 1
Cerebral artery stenosis (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Early satiety (General disorders) | 0 | 1
Gait disturbance (General disorders) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Sinus arrest (Cardiac disorders) | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 1
Aortic thrombosis (Vascular disorders) | 0 | 1
Intermittent claudication (Vascular disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Colon operation (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Xeomin Short Flex (N=142) | Xeomin Long Flex (N=140)
Dysphagia (Gastrointestinal disorders) | 36 | 35
Headache (Nervous system disorders) | 12 | 17
Muscular weakness (Musculoskeletal and connective tissue disorders) | 10 | 12
Neck pain (Musculoskeletal and connective tissue disorders) | 9 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 10
Fall (Injury, poisoning and procedural complications) | 8 | 7
Nausea (Gastrointestinal disorders) | 6 | 9
Sinusitis (Infections and infestations) | 6 | 7
Upper respiratory tract infection (Infections and infestations) | 9 | 4
Dizziness (Nervous system disorders) | 5 | 7
Nasopharyngitis (Infections and infestations) | 8 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.